CLINICAL TRIAL: NCT00668408
Title: Long-Term Oxygen Therapy (LTOT) in Chronic Obstructive Pulmonary Disease (COPD) Patients With Moderate Chronic Hypoxemia and Chronic Heart Failure (CHF)
Brief Title: LTOT in COPD Patients With Moderate Chronic Hypoxemia and Chronic Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Antonio Corrado, Azienda Ospedaliero-Universitaria Careggi Firenze (UTIP)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM6YHYW4
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Lung Diseases, Obstructive; Chronic Heart Failure; Chronic Hypoxemia
Keywords: OTLT; COPD; CHRONIC HYPOXEMIA; CHF
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Oxygen; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LTOT group (Other): Study group: optimal medical therapy plus LTOT = or > 15 hours pro die
  Interventions: Other: LTOT (oxygen therapy)
- Non LTOT group (Other): control group: optimal medical therapy without LTOT
  Interventions: Other: Pharmacological therapy of COPD and CHF

INTERVENTIONS:
Other: LTOT (oxygen therapy) — Patients on LTOT will receive oxygen for at least 15 hours/day from the liquid oxygen systems at a flow rate adjusted to raise resting SaO2 between 93 and 96% and / or PaO2 between 65 and 80 mmHg every day for 3 years.
  Other Names: LTOT treatment
  Arms: LTOT group
Other: Pharmacological therapy of COPD and CHF — Optimal pharmacologic treatment will include :
  * Long (LABD, salmeterol, formoterol, tiotropium) - as well as short-acting (SABD, Salbutamol, terbutaline, ipratropium)bronchodilators (beta-2 agonists, anticholinergics)
  * Inhaled steroids (ICS, beclomethasone, fluticasone, budesonide always associated with LABD)
  * Beta-blockers
  * Diuretics
  * Angiotensin-converting enzyme (ACE) inhibitors alone or in associations with diuretics
  * Statins and any other treatment required for associated co-morbidities (eg insulin and/or anti-diabetic drugs, other antihypertensive, etc).
  The treatment of the deseases will follow the international guidelines.
  Other Names: Pharmacological treatment
  Arms: Non LTOT group

SUMMARY:
In patients with both COPD and CHF, moderate chronic hypoxemia is caused by a combination of intrapulmonary and extrapulmonary factors. The hypothesis of this study is that adequate medical therapy for both conditions can correct the moderate hypoxemia by improving the underlying mechanisms without the need of LTOT. If this hypothesis is correct, the study will provide a valuable information to the Italian Agency of drugs (Agenzia Italiana del Farmaco, AIFA) to reduce the inappropriate use of LTOT for COPD patients with moderate hypoxemia and CHF, and will help the Italian National Health Service to reduce both the direct and indirect costs of unnecessary LTOT.

DETAILED DESCRIPTION:
Long-term oxygen treatment (LTOT) improves survival of COPD patients with severe hypoxemia . The improved survival was proven in COPD patients with severe chronic hypoxemia (PaO2< or = 55 mmHg), providing oxygen was delivered for = or >15 hours/day. Since then, > 15 hours/day LTOT has become the standard treatment for COPD patients with severe hypoxemia. LTOT has been extended without evidence to COPD patients with moderate hypoxemia (55< PaO2 <60mmHg), when associated with some clinical and laboratory signs of cardiac diseases and to patients with decreased oxygen saturation (SO2 < 90%) during exercise or sleep. Chronic heart failure (CHF) is a common co-morbidity of COPD (>30% ) particularly in the elderly. Whether LTOT improves survival in patients with moderate chronic hypoxemia and CHF is unknown. This is an issue of concern because of the potential importance of LTOT in severe COPD, and of the cost of LTOT (about Euro 250 millions/year in Italy). The aim of this 3 year randomized clinical trial is to investigate whether, in COPD patients with moderate hypoxemia associated with CHF treatment including LTOT is no different from treatment without LTOT in term of survival and of exacerbations, hospitalizations, and quality of life. The study will be conducted in 76 Italian hospital pulmonary units, and will start on May 15th 2008 and end on October 31st 2012. One thousand stable COPD patients treated according to COPD and CHF international guidelines will be randomized to treatment including LTOT (Study Group) or treatment without LTOT (Control Group). All patients will regularly undergo clinical assessment, arterial blood gases (3 monthly), and Saint George's Respiratory Questionnaire (SGRQ, 6 monthly),and will be contacted with monthly telephone calls.

Considering 1) the lack of evidence supporting LTOT in COPD patients with moderate hypoxemia and CHF, 2) the pathophysiology of CHF , and 3) the improvement of pharmacological treatment of both COPD and CHF, we expect that, after optimization of medical therapy, LTOT will not improve survival or frequency and severity of exacerbations and/or hospitalization, and not even quality of life due to the balance of small clinical benefits (improved exercise tolerance, better sleep) with the inconveniences associated with LTOT. This non-inferiority study is powered on survival, which is the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 > 80 years
* Confirmed COPD (GOLD criteria)
* Moderate and stable hypoxemia (55< PaO2 <65 mmHg)
* Clinical signs of CHF (ESC criteria)
* Ex-smokers (> 20 pack/years) since at least 3 months

Exclusion Criteria:

* Clinical instability and/or exacerbation
* Congenital heart diseases
* Lung cancer
* Thoracic restrictive disorders
* Other coexisting diseases influencing 3-yr survival

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-05; Primary Completion 2012-03 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is mortality. | 3 years

SECONDARY OUTCOMES:
Secondary endpoint of the study is to evaluate whether the appropriate medical treatment without LTOT is not inferior to medical treatment with LTOT in terms of quality of life, rate and severity of exacerbation, number of hospital admissions. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Corrado, MD, Principal Investigator — AOU Careggi
Locations (66):
- Italy (66):
  - Ausl 8 di Arezzo, Arezzo, AR
  - Azienda Ospedaliera S. G. Moscati, Avellino, AV
  - A.O. Universitaria Ospedale consorziale policlinico di Bari, Bari, BA
  - Presidio ospedaliero Barletta, Barletta, BA
  - Azienda ospedale G. Rummo, Benevento, BN
  - Irccs Fondazione Maugeri, Gussago, BS
  - Ospedale Roberto Binaghi, Cagliari, CA
  - Presidio Ospedaliero F.lli Crobu Iglesias, Iglesias, CI
  - Asp di Cosenza - Ambito territoriale di Castrovillari (ex asl 2), Castrovillari, CS
  - Asp di Catanzaro - Ambito territoriale di catanzaro (ex asl 7), Catanzaro, CZ
  - Azienda Ospedaliera Mater Domini, Catanzaro, CZ
  - Presidio Ospedaliero Morgagni-Pierantoni di Forlì, Forlì, FC
  - Presidio Ospedaliero Morgagni-Pierantoni, Forlì, FC
  - A.O. Universitaria Arcispedale S. Anna, Ferrara, FE
  - A.O. Universitaria Careggi, Florence, FI
  - Irccs fondazione Don Gnocchi - Centro S. Maria agli ulivi, Impruneta, FI
  - A.O. Universitaria S. Martino, Genova, GE
  - Ospedale della Misericordia, Grosseto, GR
  - Ospedale S. Andrea, Massa Marittima, GR
  - Stabilimento ospedaliero di Imperia, Imperia, IM
  - Ospedale generale prov. card. G. Panico, Tricase, LE
  - Ausl 2 di Lucca, Lucca, LU
  - Ospedale S. Giuseppe f.b.f., Milan, MI
  - Ospedale civile di Vimercate, Vimercate, MI
  - Presidio Ospedaliero C. Poma, Mantova, MN
  - A.O. Universitaria policlinico di Modena, Modena, MO
  - Ospedale Civile di Carrara, Carrara, MS
  - A.O. V. Cervello, Palermo, PA
  - Presidio ospedaliero Civico e benfratelli, Palermo, PA
  - Aulss 15 alta padovana, Cittadella, PD
  - Azienda Ospedaliera di padova, Padua, PD
  - A.O. di Perugia - Ospedale S. Maria della Misericordia (ex Silvestrini), Perugia, PG
  - Asl 2 di Perugia, Perugia, PG
  - A.O. Universitaria Pisana, Pisa, PI
  - Azienda Ospedaliera S. Maria degli angeli, Pordenone, PN
  - A.O. Universitaria di Parma, Parma, PR
  - Ausl 3 di Pistoia, Pistoia, PT
  - Irccs fondazione Maugeri, Montescano, PV
  - Irccs Fondazione Maugeri, Pavia, PV
  - Irccs policlinico S. Matteo, Pavia, PV
  - Ospedale S. Sebastiano, Correggio, RE
  - Ospedale di S. Maria Nuova, Reggio Emilia, RE
  - Ospedale S. Camillo De Lellis, Rieti, RI
  - Ausl rm/h di Albano Laziale, Albano Laziale, RM
  - A.O. Universitaria Policlinico Tor Vergata, Roma, RM
  - Az. Osp. San Camillo-Forlanini, Roma, RM
  - Az.osp.san camillo-forlanini -, Roma, RM
  - Aulss 18 di Rovigo, Rovigo, RO
  - Asl sa/2 di Salerno, Salerno, SA
  - A.O. Universitaria senese, Siena, SI
  - Presidio ospedaliero San Bartolomeo, Sarzana, SP
  - Azienda Ospedaliera Umberto I, Syracuse, SR
  - A.O. Universitaria Policlinico di Sassari, Sassari, SS
  - Az. Osp. Ospedale S. Corona, Pietra Ligure, SV
  - Ospedale Mazzini, Teramo, TE
  - Ospedale di Trento - P.O. S.Chiara, Trento, TN
  - A.O. Universitaria S. Giovanni Battista-Molinette di Torino, Torino, TO
  - A.O. Universitaria ospedali riuniti di Trieste, Trieste, TS
  - Ospedale di, Vicenza, VI
  - Ospedale civile Orlandi Bussolengo, Bussolengo, VR
  - Terapia Intensiva Pneumologica- AOU Careggi, Florence
  - Azienda ospedaliera "A. Cardarelli", Napoli
  - Azienda Ospedaliera Antonio Cardarelli di Napoli, Napoli
  - Azienda Ospedaliera Cotugno, Napoli
  - A.O. Universitaria Maggiore della Carità, Novara
  - Irccs Fondazione Maugeri, Veruno